CLINICAL TRIAL: NCT05104892
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, 12 Week Proof-of-Concept (PoC) Study to Assess the Efficacy, Safety, and Tolerability of Rilzabrutinib in Participants With Moderate-to-severe Asthma Who Are Not Well Controlled on Inhaled Corticosteroid (ICS) Plus Long-acting β2 Adrenergic Agonist (LABA) Therapy
Brief Title: Proof of Concept Study of Rilzabrutinib in Adult Participants With Moderate-to-severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17208; U1111-1262-2956 (Registry Identifier: ICTRP); 2021-002490-26 (EudraCT Number)
Record Dates: First submitted 2021-10-17; First posted 2021-11-03 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rilzabrutinib (Experimental): Rilzabrutinib BID or TID and ICS/LABA
  Interventions: Drug: Rilzabrutinib
- Placebo (Placebo Comparator): Placebo and ICS/LABA
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rilzabrutinib — Pharmaceutical form: Tablet Route of administration: Oral
  Other Names: PRN1008/SAR444671
  Arms: Rilzabrutinib
Drug: placebo — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
This is a parallel, treatment, Phase 2, double-blind, 2 arm, 12-week Proof of Concept (PoC) study with 2 staggered cohorts (2 arms in each cohort) that is designed to assess the efficacy, safety, and tolerability of rilzabrutinib in adult participants (aged 18-70 years) with moderate-to-severe asthma who are not well controlled on ICS/LABA therapy. Study treatment includes investigational medicinal product (IMP) (rilzabrutinib or placebo) added-on to a background therapy of ICS/LABA (fluticasone/salmeterol [non-investigational medicinal product], standardized at screening). Background therapy of ICS/LABA will be withdrawn during the 12week randomized treatment period and resumed at the end of the IMP treatment period, as outlined below:

* Screening period (4 weeks)
* Randomized IMP treatment period (12 weeks ± 3 days)

  * Background therapy stabilization phase (4 weeks)
  * Background therapy withdrawal phase (4-5 weeks)
  * No background therapy phase (3-4 weeks)
* Post IMP treatment safety follow-up period (4 weeks ± 3 days)

DETAILED DESCRIPTION:
The total study duration per participant is expected to be up to 20 weeks: up to 4 weeks screening, 12 weeks on-treatment double-blind period, and 4-week post-IMP treatment follow up.

ELIGIBILITY:
Inclusion Criteria:

* A physician diagnosis of asthma for at least 12 months based on the Global Initiative for Asthma (GINA) 2018,2019, 2020 Guidelines.
* Participants with existing treatment with at least moderate to high doses of ICS therapy in combination with a LABA as second controller for at least 3 months with a stable dose ≥1 month prior to Visit 1.
* Participants with prebronchodilator FEV1 >40% of predicted normal at Visit 1/Screening. Prebronchodilator FEV1 ≥50% of predicted normal at Visit 2/Baseline.
* Participants with reversibility of at least 12% and 200 mL in FEV1 15 to 30 minutes after administration of 2 to 4 puffs (200-400 mcg) of albuterol/salbutamol or levalbuterol/levosalbutamol during screening or documented history of a reversibility test that meets this criterion within 5 years prior to Visit 1 or documented positive response to methacholine challenge (a decrease in FEV by 20% [PC20] of <8mg/mL) within 5 years prior to Visit 1/Screening is considered acceptable to meet this inclusion criterion.
* Participants must have experienced, within 2 years prior to Visit 1, any of the following asthma exacerbation events at least once: Treatment with a systemic steroid (oral or parenteral) for worsening asthma OR Hospitalization or emergency medical care visit for worsening asthma.
* Body mass index (BMI) ≥17.5 and ≤40 kg/m2
* All Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Participants must have completed COVID-19 vaccination per current regional health authority recommendations prior to screening.

Exclusion Criteria:

* History of serious infections requiring intravenous therapy with the potential for recurrence (as judged by Site Investigator), with less than 4 weeks interval between resolution of serious infection and first dose of study drug, or currently active moderate-to-severe infection at Screening (Grade 2 or higher).
* Chronic lung disease (for example, chronic obstructive pulmonary disease [COPD], or idiopathic pulmonary fibrosis [IPF]) which may impair lung function, or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts, for e.g. eosinophilic granulomatosis with polyangiitis.
* History of life-threatening asthma (i.e., severe exacerbation that requires intubation).
* Participants with any of the following events within the 4 weeks prior to their Screening Visit 1 or during the screening period: Treatment with 1 or more systemic (oral and/or parenteral) steroid bursts for worsening asthma OR Hospitalization or emergency medical care visit for worsening asthma
* Asthma Control Questionnaire 5-question version (ACQ-5) score <1.25 or >3.0 at V2/randomization. During the screening period an ACQ-5 of up to ≤4 is acceptable.
* Current smoker or cessation of smoking within the 6 months prior to Visit 1.
* Previous smoker with a smoking history >10 pack-years.
* Current or chronic history of liver disease.
* Known hepatic or biliary abnormalities, e.g. moderate or severe hepatic impairment, such as Child Pugh B or C
* Symptomatic herpes zoster within 3 months prior to screening.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate rilzabrutinib/placebo absorption.
* Conditions that may predispose the participant to excessive bleeding
* History of solid organ transplant.
* A history of malignancy of any type within 5 years before Day 1, other than surgically excised non-melanoma skin cancers or in situ cervical cancer.
* Is not up-to-date with recommended vaccinations per local guidelines.
* Anti-immunoglobulin E (IgE) therapy (e.g., omalizumab [Xolair®]) within 130 days prior to Visit 1 or any other biologic therapy (including anti-IL4/4R or IL-5/5R monoclonal antibodies [mAb]) or systemic immunosuppressant (e.g., methotrexate) to treat inflammatory disease or autoimmune disease (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis) and other diseases, within 2 months or 5 half-lives prior to Visit 1, whichever is longer.
* Use of inhalers other than ICSs, LABAs, and short-acting beta agonists (no long-acting muscarinic antagonists (LAMAs) or mucolytics) and leukotriene receptor antagonists (montelukast, zafirkulast) during the study period.
* Participants who have received bronchial thermoplasty within 2 years prior to Visit 1 or plan to begin therapy during the screening period or the randomized treatment period.
* Use of proton pump inhibitor drugs such as omeprazole and esomeprazole within 3 days of Day 1.
* Use of known systemic strong-to-moderate inducers or inhibitors of CYP3A within 14 days or 5 half-lives (whichever is longer) of Study Day 1 and until the end of the active treatment period.
* Live vaccine except Bacille Calmette Guerinn-vaccination within 28 days prior to Day 1 or plans to receive one during the trial; Calmette Guerin-vaccination within 12 months prior to Screening.
* COVID-19 vaccine within 14 days prior to Study Day 1.
* Previous use of a Bruton tyrosine kinase (BTK) inhibitor.
* Has received any investigational drug (or is currently using an investigational device) within the 30 days before Day 1, or at least 5 times the respective elimination half-life time (whichever is longer).
* Electrocardiogram (ECG) findings of QT corrected for heart rate (QTc) >450 msec (males) or >470 msec (females), poorly controlled atrial fibrillation (i.e., symptomatic patients or a ventricular rate above 100 beats/min on ECG), or other clinically significant cardiovascular abnormalities.
* Active COVID-19 infection as documented by a positive COVID-19 molecular test.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an LOAC event during the treatment period | Until Week 12
  Loss of Asthma Control (LOAC) event is defined as any of the following:
  * A 30% or greater reduction from baseline in morning peak expiratory flow (PEF) on 2 consecutive days
  * ≥6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days
  * Increase in ICS ≥4 times the last prescribed ICS dose (or ≥50% of the prescribed ICS dose at V2 if background therapy withdrawal completed)
  * Requiring use of systemic (oral and/or parenteral) steroid treatment
  * Requiring hospitalization or emergency room visit for asthma exacerbation

SECONDARY OUTCOMES:
Pre-bronchodilator FEV1 (Forced expiratory volume in one second) change from baseline to EOT (end of treatment) | From baseline to Week 12
Post-bronchodilator FEV1 change from baseline to EOT | From baseline to Week 12
The absolute change in the percent predicted FEV1 from baseline to EOT (pre- and post-bronchodilator) | From baseline to Week 12
Change from baseline in pre- and post-bronchodilator FEV1 and forced vital capacity [FVC] at each spirometry endpoint | From baseline until Week 12
Change from baseline in peak expiratory flow [PEF] and forced expiratory flow [FEF] 25-75% at each spirometry endpoint | From baseline until Week 12
Asthma Control Questionnaire-5 (ACQ-5) score change from baseline at EOT and at each assessment time point | From baseline until Week 12
  The ACQ-5 is a questionnaire that measures the adequacy of asthma control and any changes in asthma control that may occur spontaneously or as a result of treatment. The ACQ-5 has five questions on the asthma symptoms and patients are asked to recall how their asthma has been during the previous week and to respond on a 7-point scale for each question (0 = no impairment, 6 = maximum impairment). The ACQ-5 score is the mean of the 5 questions and, therefore, between 0 (totally controlled) and 6 (severely uncontrolled). A high score indicates low asthma control.
Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ[S]) Self-administered score change from baseline at EOT and at each assessment time point | From baseline until Week 12
  The AQLQ(S) was designed as a self-administered patient reported outcome to measure the functional impairments that are most troublesome to adolescents and adults ≥12 years of age as a result of their asthma. The instrument is comprised of 32 items, each rated on a 7-point Likert scales from 1 to 7. Higher scores indicate better quality of life.
Change in Asthma Daytime Symptom Diary (ADSD) and Asthma Nighttime Symptom Diary (ANSD) scores from baseline to EOT and each week | From baseline until Week 12
  ADSD and ANSD assess asthma severity based on patient self-report of asthma core symptoms, i.e., difficulty of breathing; wheezing; shortness of breath; chest tightness; chest pain; and cough. Both the ADSD and ANSD are composed of 6 items rated using an 11-point numerical rating scale (NRS) that ranges from 0 = None to 10 = As bad as you can imagine. The participants will record their daytime and nighttime asthma symptoms in an electronic diary, once in the evening and once in the morning, respectively.
Plasma pharmacokinetic (PK) concentrations of rilzabrutinib in participants with asthma | Until Week 16
Participants with Treatment Emergent Adverse Events | Until Week 16
Change in numbers of inhalations/day of albuterol or levalbuterol for symptom relief from baseline to EOT and each week | From baseline until Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (51):
- Argentina (6):
  - Investigational Site Number : 0320004, Berazategui, Buenos Aires
  - Investigational Site Number : 0320006, CABA, Buenos Aires
  - Investigational Site Number : 0320003, CABA, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320005, Ciudad Autonoma Buenos Aires
  - Investigational Site Number : 0320002, Ciudad Autonoma Buenos Aires
- Bulgaria (4):
  - Investigational Site Number : 1000004, Kozloduy
  - Investigational Site Number : 1000001, Rousse
  - Investigational Site Number : 1000003, Sevlievo
  - Investigational Site Number : 1000002, Sofia
- Canada (2):
  - Investigational Site Number : 1240006, Vancouver, British Columbia
  - Investigational Site Number : 1240005, Waterloo, Ontario
- Chile (7):
  - Investigational Site Number : 1520005, Curicó, Maule Region
  - Investigational Site Number : 1520002, Talca, Maule Region
  - Investigational Site Number : 1520007, Santaigo, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Quillota, Región de Valparaíso
- Investigational Site Number : 6420001, Düsseldorf, Germany
- Hungary (3):
  - Investigational Site Number : 3480001, Edelény
  - Investigational Site Number : 3480004, Hajdunánás
  - Investigational Site Number : 3480003, Pécs
- Mexico (5):
  - Investigational Site Number : 4840001, Guadalajara, Jalisco
  - Investigational Site Number : 4840002, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, San Juan del Río, Querétaro
  - Investigational Site Number : 4840003, Durango
  - Investigational Site Number : 4840004, Veracruz
- Poland (9):
  - Investigational Site Number : 6160009, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160007, Lublin, Lubusz Voivodeship
  - Investigational Site Number : 6160003, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160006, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160005, Bialystok
  - Investigational Site Number : 6160002, Krakow
  - Investigational Site Number : 6160010, Lodz
  - Investigational Site Number : 6160001, Lodz
  - Investigational Site Number : 6160008, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Investigational Site Number : 6420002, Cluj-Napoca, Romania
- South Korea (6):
  - Investigational Site Number : 4100007, Daegu, Daegu
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul
- Spain (3):
  - Investigational Site Number : 7240004, Santander, Cantabria
  - Investigational Site Number : 7240003, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Málaga
- Turkey (Türkiye) (2):
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920001, Mersin
- United Kingdom (2):
  - Investigational Site Number : 8260002, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260001, Bradford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371